CLINICAL TRIAL: NCT00002618
Title: A Phase III Study of Large Cell Lymphomas in Children and Adolescents: Comparison of APO vs APO + IDMTX/HDARA-C and Continuous vs Bolus Infusion of Doxorubicin
Brief Title: Combination Chemotherapy in Treating Pediatric Patients With Advanced-Stage Large Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 9315; POG-9315 (Other: Pediatric Oncology Group); CDR0000063955 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating | interventions — Filgrastim; pegfilgrastim; Granulocyte Colony-Stimulating Factor; Cytarabine; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (Active Comparator): Patients begin radiotherapy (5 days a week for 4.5 weeks) to residual tumor on day 1 of maintenance.
  Interventions: Biological: filgrastim; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy
- Regimen B (Active Comparator): Patients receive whole brain irradiation (5 days a week for 3.1 weeks) beginning on day 1 of maintenance. Patients are followed monthly for 6 months, every 3 months for 18 months, every 6 months for 3 years, and annually thereafter.
  Interventions: Biological: filgrastim; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: rmetHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: cytarabine
  Other Names: CYTOSINE ARABINOSIDE; Ara-C; Cytosar; NSC #63878
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127
Drug: leucovorin calcium
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #3590
Drug: mercaptopurine
  Other Names: 6-MP; Purinethol; NSC #755
Drug: methotrexate
  Other Names: amethopterin; NSC #740
Drug: prednisone
  Other Names: Deltasone; Meticorten; Liquid Pred; NSC #10023
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #67574
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Giving the drugs in different doses may kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy with various combinations of drugs in treating pediatric patients with advanced-stage large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the event free survival of children with advanced stage large cell lymphoma treated with modified APO (doxorubicin/prednisone/vincristine/mercaptopurine) with or without intermediate-dose methotrexate/high dose cytarabine as maintenance therapy following induction therapy with APO. II. Characterize further the immunophenotypic and morphologic correlates of pediatric large cell lymphoma.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms, except for those with CNS disease. These patients are assigned to arm II and receive whole brain irradiation on Regimen B. Arm I: Induction (Modified APO): Patients receive vincristine IV on days 1, 8, 15, 22, and 29, doxorubicin IV over 15 minutes on days 1 and 22, prednisone three times a day on days 1-28, and methotrexate intrathecally (IT) on days 1, 8, and 22. Patients in complete remission on day 43 proceed to maintenance, those in partial remission undergo biopsy then proceed to maintenance, and those with residual disease receive radiotherapy on regimen A concurrently with maintenance. Maintenance (day 1 is day 43 of Induction): Courses of intermediate dose methotrexate/leucovorin calcium and high dose cytarabine (ID MTX/CF/HD ARA-C) and modified APO alternate every 3 weeks. Patients receive a total of 15 courses (8 of ID MTX/CF/HD ARA-C and 7 of Modified APO). ID MTX/CF/HD ARA-C: Patients receive methotrexate IV over 24 hours on day 1, leucovorin calcium IV or orally every 6 hours on days 2 and 3, cytarabine IV over 48 hours on days 2 to 4, and methotrexate IT on day 1 of courses 1, 3, and 5. Filgrastim (G-CSF) is administered beginning on day 5 and continuing until blood counts recover. Modified APO: Patients receive vincristine IV on day 1, oral mercaptopurine on days 1-5, doxorubicin IV over 15 minutes on day 1, and oral prednisone three times a day on days 1-5. Arm II: Induction: Patients receive treatment as in arm I except that patients with CNS disease also receive methotrexate IT on days 15, 29, and 36. Maintenance (day 1 is day 43 of Induction): Modified APO: as in Arm I, with methotrexate administered on day 1 of courses 1, 3, and 5 (days 1-5 for patients with CNS disease). Courses repeat every 21 days for a total of 15 courses. Patients with CNS disease begin radiotherapy on Regimen B on week 2 of maintenance. Regimen A: Patients begin radiotherapy (5 days a week for 4.5 weeks) to residual tumor on day 1 of maintenance. Regimen B: Patients receive whole brain irradiation (5 days a week for 3.1 weeks) beginning on day 1 of maintenance. Patients are followed monthly for 6 months, every 3 months for 18 months, every 6 months for 3 years, and annually thereafter.

PROJECTED ACCRUAL: A total of 242 patients will be accrued for this study over approximately 5.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated large cell lymphoma, including the following histologic designations: Rappaport classification Diffuse histiocytic Mixed lymphocytic-histiocytic Working Formulation classification Diffuse large cell, cleaved and/or noncleaved Immunoblastic Diffuse, mixed small and large cell Lukes-Collins classification Diffuse large cleaved Diffuse large noncleaved Immunoblastic T or B cell True histiocytic Updated Kiel classification Cytocentric large cell Centroblastic-centrocytic T-zone Lymphoepithelioid cell (Lennert's) Immunoblastic T or B cell Large cell anaplastic Pleomorphic Centroblastic-centrocytic, diffuse Malignant histiocytosis Murphy stage III/IV HIV-associated lymphoma eligible Any degree of bone marrow involvement eligible CNS disease eligible (such patients not randomized)

PATIENT CHARACTERISTICS: Age: Under 22 Performance status: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No prior therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 242 (Estimated)
Dates: Start 1994-12; Primary Completion 2000-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Event free survival | Length of study
  To study whether intermediate-dose methotrexate/high-dose Ara-C (ID MTX/HDAra-C), administered during the maintenance phase can improve the event free survival (EFS) of patients with advanced-stage large cell lymphoma (LCL).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Laver, MD, Study Chair — Medical University of South Carolina
Locations (10):
- United States (8):
  - Via Christi Regional Medical Center-Saint Francis Campus, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Memorial Mission Hospital, Asheville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland

REFERENCES:
- [Background] Hutchison RE, Laver JH, Chang M, Muzzafar T, Desai S, Murphy S, Schwenn M, Shuster J, Link MP; Children's Oncology Group. Non-anaplastic peripheral t-cell lymphoma in childhood and adolescence: a Children's Oncology Group study. Pediatr Blood Cancer. 2008 Jul;51(1):29-33. doi: 10.1002/pbc.21543. PMID 18300314
- [Background] Hutchison RE, Finch C, Kepner J, Fuller C, Bowman P, Link M, Schwenn M, Laver J, Desai S, Barrett D, Murphy SB. Burkitt lymphoma is immunophenotypically different from Burkitt-like lymphoma in young persons. Ann Oncol. 2000;11 Suppl 1:35-8. PMID 10707776
- [Result] Nasr MR, Laver JH, Chang M, Hutchison RE. Expression of anaplastic lymphoma kinase, tyrosine-phosphorylated STAT3, and associated factors in pediatric anaplastic large cell lymphoma: A report from the children's oncology group. Am J Clin Pathol. 2007 May;127(5):770-8. doi: 10.1309/FNY8Y4H6PK1V2MGE. PMID 17439836
- [Result] Laver JH, Kraveka JM, Hutchison RE, Chang M, Kepner J, Schwenn M, Tarbell N, Desai S, Weitzman S, Weinstein HJ, Murphy SB. Advanced-stage large-cell lymphoma in children and adolescents: results of a randomized trial incorporating intermediate-dose methotrexate and high-dose cytarabine in the maintenance phase of the APO regimen: a Pediatric Oncology Group phase III trial. J Clin Oncol. 2005 Jan 20;23(3):541-7. doi: 10.1200/JCO.2005.11.075. PMID 15659500